CLINICAL TRIAL: NCT06650423
Title: ONCO-ADHER: Adherence to Treatment With a Aromatase Inhibitors With or Without Abemaciclib in Patients With Early-stage, Endocrine-dependent, HER-2-negative Breast Cancer
Brief Title: Adherence to Aromatase Inhibitors ± Abemaciclib Treatment in Patients With Early-stage HER2-negative Breast Cancer
Acronym: ONCO-Adher
Status: Not yet recruiting | Type: Observational
Sponsor: Erika Matos (Other)
Collaborators: University of Ljubljana (Other)
Responsible Party: Sponsor-Investigator, Erika Matos, assoc. prof. Erika Matos, MD, PhD, Institute of Oncology Ljubljana
Organization: Institute of Oncology Ljubljana (Other)
Other Study IDs: ORI2024-001
Record Dates: First submitted 2024-10-16; First posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Early Breast Cancer; Hormone Receptor Positive Tumor; HER2-negative Breast Cancer
Keywords: breast cancer; medication adherence; CDK4/6; HR+; HER2-; aromatase inhibitor; quality of life; medication belief
MeSH Terms: conditions — Breast Neoplasms; Medication Adherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Aromatase inhibitor + abemaciclib: Adult women with early HR+ HER2- breast cancer, eligible for treatment with aromatase inhibitor + abemaciclib, both prescribed prior inclusion into study, irrespective of protocol, as per regular clinical practice
- Aromatase inhibitor: Adult women with early HR+ HER2- breast cancer, eligible for treatment with aromatase inhibitor, prescribed prior inclusion into study, irrespective of protocol, as per regular clinical practice

SUMMARY:
Around 90% of breast cancer patients are diagnosed at an early stage and approximately 70%, are hormone receptor-positive and HER2-negative (HR+/HER2-). Despite advancements in adjuvant endocrine therapy, 20-30 % of early-stage BC patients relapse within the first decade post-surgery. Recent clinically meaningful therapeutic option for these patients has been cyclin-dependent kinases 4/6 inhibitors (CDK4/6 inhibitors). Abemaciclib and ribociclib, were assessed in the adjuvant setting, both showing improvement in IDFS. Abemaciclib has been approved by the FDA and EMA for HR+/HER2- early breast cancer at high risk of disease recurrence and is the first addition to Slovenian treatment regimen in routine clinical practice. Poor medication adherence can directly affect the effectiveness of treatment for early HR+/HER2- breast cancer. While adherence data in patients treated with aromatase inhibitors are available, the adherence rate in patients with early HR+/HER2- breast cancer taking abemaciclib is unclear. In this study, investigators hypothesize that patients receiving abemaciclib in combination with aromatase inhibitors will have a lower medication adherence and higher discontinuation rate compared to those receiving aromatase inhibitors alone. It is expected that patient with better quality of life, cognitive functioning and more positive attitude towards their therapy will demonstrate higher medication adherence rate. Adherence rate will also be affected by other factors, such as age and prior treatments.

DETAILED DESCRIPTION:
Breast cancer (BC) is the most prevalent malignant tumour in women, with an estimated 2.308 million new cases and over 665,000 deaths globally in 2022. Around 90% of patients are diagnosed at an early stage and the majority of these cases, approximately 70%, are hormone receptor-positive and HER2-negative (HR+/HER2-). Despite advancements in adjuvant endocrine therapy that significantly lower recurrence and mortality rates, 20-30 % of early-stage BC patients experience relapse within the first decade post-surgery. Around 12% of patients with HR+/HER2- BC belong to high-risk population with 5-years invasive disease-free survival (IDFS) of 70.2% vs 90.0% in non-high-risk. The most recent clinically meaningful therapeutic option for these patients has been cyclin-dependent kinases 4/6 inhibitors (CDK4/6 inhibitors). Endocrine therapy combined with CDK4/6 inhibitors (abemaciclib, palbociclib, and ribociclib) is now the standard, most effective, and recommended treatment for these patients in the first or subsequent lines of treatment for advanced disease. Two CDK4/6 inhibitors, abemaciclib and ribociclib, have been assessed also for use in the adjuvant setting (MonarchE and NATALEE study). Both studies showed improvement in IDFS of combined endocrine therapy and CDK4/6 inhibitor vs endocrine therapy alone. Abemaciclib has been approved by both the FDA and EMA for patients with HR+/HER2- early breast cancer at high risk of disease recurrence and has therefore recently been added to Slovenian current regimen for this indication in routine clinical practice. Non-adherence to adjuvant therapy may compromise the efficacy of combined treatment in preventing disease recurrence and mortality. Some historical data report that only 60-70% of patients with early BC adhere to adjuvant therapy, making adherence a significant challenge. Key factors influencing adherence to cancer treatment include the perceived benefits of the treatment, the setting in which the treatment is administered (at home or in a hospital), the associated risks, the impact on quality of life, and the costs involved. Non-adherence often arises because patients do not experience the immediate benefits. With no visible or measurable signs of the disease and no physical symptoms of the disease, as is the case in patients receiving adjuvant treatment, and given that many would not have experienced a relapse even without adjuvant therapy, patients are much more likely to discontinue treatment if they experience adverse events/reactions (AE). Adherence to treatment with CDK4/6 inhibitors in combination with aromatase inhibitors differs from some other systemic treatments due to the continuous treatment regimen that lasts for several years without interruption. In early BC, it lasts two (abemaciclib) or three (ribociclib) years and is associated with some specific AEs. Aromatase inhibitors are associated with arthralgias, myalgias, and joint stiffness, whereas CDK4/6 inhibitors with myelotoxicity, hepatotoxicity and gastrointestinal symptoms (especially diarrhoea caused by abemaciclib). The duration of treatment, five or more vs two years (aromatase inhibitors as monotherapy vs abemaciclib in combination with aromatase inhibitors, respectively), may lead to different discontinuation rates. Despite the growing amount of real-world experiences with combined treatment with aromatase inhibitors and abemaciclib in the adjuvant setting, there is currently a lack of literature specifically exploring how patient adherence and attitudes are influenced by this combination. This gap underscores the need for further research to fully understand the impact of these therapies on medication adherence. Poor medication adherence can directly affect the effectiveness of treatment for early HR+/HER2- breast cancer. While data on medication adherence in patients taking aromatase inhibitors are available, the adherence rate in patients with early HR+/HER2- breast cancer taking abemaciclib remains unclear. Due to the differing characteristics of these treatment modalities, particularly their distinct safety profiles, medication adherence and persistence may vary between them. It is hypothesized that patients receiving abemaciclib in combination with aromatase inhibitors will have a lower medication adherence and higher discontinuation rate compared to those receiving aromatase inhibitors alone. It's also expected that patient with better quality of life, better cognitive functioning and more positive attitude towards their therapy will demonstrate higher medication adherence rate. Additionally, it's anticipated that other factors, such as age and prior treatments, will also contribute to adherence rates.

ELIGIBILITY:
Inclusion Criteria:

* Female,
* Early HR+/HER-2- BC,
* Patient is receiving adjuvant therapy with an aromatase inhibitor (letrozole, anastrozole or exemestane), with or without a CDK4/6 inhibitor abemaciclib, for no more than 18 months,
* Treatment of BC is being conducted at OIL,
* Patient has mandatory health insurance through Health Insurance Institute of Slovenia,
* Patient understands Slovenian language, and
* Patient agrees to participate in the study and provides written informed consent.

Exclusion Criteria:

* Metastatic HR+/HER-2- BC
* Previous treatment for BC with an aromatase inhibitor, with or without a CDK4/6 inhibitor, due to BC.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Adult women, sex at birth female
Study Population: Eligible adult women with early HR+ HER2- breast cancer patients.
Sampling Method: Non-Probability Sample
Enrollment: 319 (Estimated)
Dates: Start 2024-10-20 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Medication adherence in proportion of days covered (PDC) | Month 3 after starting dose
  The primary aim of this study is to determine medication adherence among HR+/HER2- early BC patients undergoing adjuvant therapy with aromatase inhibitors, either alone or in combination with abemaciclib. Medication adherence will be assessed using a combination of Medication Adherence Report Scale (MARS-5), "missed dose" questions and pill count data expressed in Proportion of Days Covered (PDC). MARS-5 scale is a self-reported questionnaire scaling from 1-5 (1=always forget, to 5=never forget) addressing non-adherence behaviors, where higher scores indicate better adherence (25 points suggests full adherence). Those with a PDC of 80% or higher will be classified as adherent, while those with a PDC below 80% will be classified as non-adherent.
Medication adherence in proportion of days covered (PDC) | Month 6 after starting dose
  The primary aim of this study is to determine medication adherence among HR+/HER2- early BC patients undergoing adjuvant therapy with aromatase inhibitors, either alone or in combination with abemaciclib. Medication adherence will be assessed using a combination of Medication Adherence Report Scale (MARS-5), "missed dose" questions and pill count data expressed in Proportion of Days Covered (PDC). MARS-5 scale is a self-reported questionnaire scaling from 1-5 (1=always forget, to 5=never forget) addressing non-adherence behaviors, where higher scores indicate better adherence (25 points suggests full adherence). Those with a PDC of 80% or higher will be classified as adherent, while those with a PDC below 80% will be classified as non-adherent.

SECONDARY OUTCOMES:
Quality of life, assessed with QLQ-C30, affecting medication adherence | Baseline visit
  Secondary aim to explore how quality of life (QoL) measured by EORTC QLQ-C30, impacts medication adherence. QLQ-C30 is a questionnaire of 30 questions (functional scales, symptom scales, single-item measures and global health status) converted into 0-100 scale. For functional and global scales, higher scores reflect better functioning or quality of life (score >70 may indicate good functioning, <70 indicating impaired functioning), whereas higher score in symptom scale represents greater severity of symptoms (>30 typically considered clinically significant, indicating notable symptom burden, <30 suggest mild or manageable symptoms). A change in 10 points or more is generally regarded as clinically meaningful change.
Quality of life, assessed with QLQ-C30, affecting medication adherence | Month 3
  Secondary aim to explore how quality of life (QoL) measured by EORTC QLQ-C30, impacts medication adherence. QLQ-C30 is a questionnaire of 30 questions (functional scales, symptom scales, single-item measures and global health status) converted into 0-100 scale. For functional and global scales, higher scores reflect better functioning or quality of life (score >70 may indicate good functioning, <70 indicating impaired functioning), whereas higher score in symptom scale represents greater severity of symptoms (>30 typically considered clinically significant, indicating notable symptom burden, <30 suggest mild or manageable symptoms). A change in 10 points or more is generally regarded as clinically meaningful change.
Quality of life, assessed with QLQ-C30, affecting medication adherence | Month 6
  Secondary aim to explore how quality of life (QoL) measured by EORTC QLQ-C30, impacts medication adherence. QLQ-C30 is a questionnaire of 30 questions (functional scales, symptom scales, single-item measures and global health status) converted into 0-100 scale. For functional and global scales, higher scores reflect better functioning or quality of life (score >70 may indicate good functioning, <70 indicating impaired functioning), whereas higher score in symptom scale represents greater severity of symptoms (>30 typically considered clinically significant, indicating notable symptom burden, <30 suggest mild or manageable symptoms). A change in 10 points or more is generally regarded as clinically meaningful change.
Quality of life, assessed with QLQ-BR23, affecting medication adherence | Baseline visit
  Secondary aim to explore how quality of life (QoL) measured by QLQ-BR23 (breast cancer specific module) questionnaire impacts medication adherence. QLQ-BR23 is a 23 question set (functional and symptom scales), transformed into 0-100 scale where higher scores in functional scales attest for better functioning whereas higher scores in symptom scales indicate greater symptom burden. For functional and global scales, higher scores reflect better functioning or quality of life (score >70 may indicate good functioning, <70 indicating impaired functioning), whereas higher score in symptom scale represents greater severity of symptoms (>20-30 typically considered clinically significant, indicating notable symptom burden).
Quality of life, assessed with QLQ-BR23, affecting medication adherence | Month 3
  Secondary aim to explore how quality of life (QoL) measured by QLQ-BR23 (breast cancer specific module) questionnaire impacts medication adherence. QLQ-BR23 is a 23 question set (functional and symptom scales), transformed into 0-100 scale where higher scores in functional scales attest for better functioning whereas higher scores in symptom scales indicate greater symptom burden. For functional and global scales, higher scores reflect better functioning or quality of life (score >70 may indicate good functioning, <70 indicating impaired functioning), whereas higher score in symptom scale represents greater severity of symptoms (>20-30 typically considered clinically significant, indicating notable symptom burden).
Quality of life, assessed with QLQ-BR23, affecting medication adherence | Month 6
  Secondary aim to explore how quality of life (QoL) measured by QLQ-BR23 (breast cancer specific module) questionnaire impacts medication adherence. QLQ-BR23 is a 23 question set (functional and symptom scales), transformed into 0-100 scale where higher scores in functional scales attest for better functioning whereas higher scores in symptom scales indicate greater symptom burden. For functional and global scales, higher scores reflect better functioning or quality of life (score >70 may indicate good functioning, <70 indicating impaired functioning), whereas higher score in symptom scale represents greater severity of symptoms (>20-30 typically considered clinically significant, indicating notable symptom burden).
Belief about medications affecting medication adherence | Baseline visit
  Secondary aim to explore how beliefs about medicines (Beliefs about medicines questionnaire- BMQ) impacts medication adherence. BMQ consists of specific and general scale, each item rated on 5-point Likers scale ranging from 1-5 (1=strongly agree, 5= strongly disagree) summing into a total score. Higher scores on specific necessity scale suggest patients strongly believe medication is essential for maintaining their health. Higher score on concerns scale indicate patients concern about medication's negative aspect, potentially leading to lowed adherence. High scores in general harm and overuse scales reflect strong beliefs in medicines in general, are harmful or overused, potentially affecting adherence.
Belief about medications affecting medication adherence | Month 3
  Secondary aim to explore how beliefs about medicines (Beliefs about medicines questionnaire- BMQ) impacts medication adherence. BMQ consists of specific and general scale, each item rated on 5-point Likers scale ranging from 1-5 (1=strongly agree, 5= strongly disagree) summing into a total score. Higher scores on specific necessity scale suggest patients strongly believe medication is essential for maintaining their health. Higher score on concerns scale indicate patients concern about medication's negative aspect, potentially leading to lowed adherence. High scores in general harm and overuse scales reflect strong beliefs in medicines in general, are harmful or overused, potentially affecting adherence.
Belief about medications affecting medication adherence | Month 6
  Secondary aim to explore how beliefs about medicines (Beliefs about medicines questionnaire- BMQ) impacts medication adherence. BMQ consists of specific and general scale, each item rated on 5-point Likers scale ranging from 1-5 (1=strongly agree, 5= strongly disagree) summing into a total score. Higher scores on specific necessity scale suggest patients strongly believe medication is essential for maintaining their health. Higher score on concerns scale indicate patients concern about medication's negative aspect, potentially leading to lowed adherence. High scores in general harm and overuse scales reflect strong beliefs in medicines in general, are harmful or overused, potentially affecting adherence.
Cognitive functioning affecting medication adherence | Baseline visit
  Secondary aim is to explore how cognitive functioning (Functinal Assessment of Cancer Therapy- Cognitive Function (FACT-Cog) impacts medication adherence. FACT-Cog consists of 37 items, divided into perceived cognitive impairments (PCI), abilities (PCA), comments form others (OTH) and impact on quality of live (QOL). Each item is scored on Likert scale from 0-4 (==never, 4=several times a day), whereas higher scores indicate better cognitive function or fewer perceived cognitive problems, higher sum of scores represent better perceived cognitive functioning.
Cognitive functioning affecting medication adherence | Month 3
  Secondary aim is to explore how cognitive functioning (Functinal Assessment of Cancer Therapy- Cognitive Function (FACT-Cog) impacts medication adherence. FACT-Cog consists of 37 items, divided into perceived cognitive impairments (PCI), abilities (PCA), comments form others (OTH) and impact on quality of live (QOL). Each item is scored on Likert scale from 0-4 (==never, 4=several times a day), whereas higher scores indicate better cognitive function or fewer perceived cognitive problems, higher sum of scores represent better perceived cognitive functioning.
Cognitive functioning affecting medication adherence | Month 6
  Secondary aim is to explore how cognitive functioning (Functinal Assessment of Cancer Therapy- Cognitive Function (FACT-Cog) impacts medication adherence. FACT-Cog consists of 37 items, divided into perceived cognitive impairments (PCI), abilities (PCA), comments form others (OTH) and impact on quality of live (QOL). Each item is scored on Likert scale from 0-4 (==never, 4=several times a day), whereas higher scores indicate better cognitive function or fewer perceived cognitive problems, higher sum of scores represent better perceived cognitive functioning.
Previous treatment affecting medication adherence | Baseline visit
  Secondary aim is to explore how factors related patient's previous treatment impact medication adherence. Previous treatment data will be gathered and descriptively presented along measured study data.
Adverse events affecting medication adherence | Baseline visit
  Secondary aim is to explore how adverse events (AE) impact medication adherence. AEs will be gathered throughout the duration of the study, assessed per seriousness, severity, causality and expectancy and descriptively presented. it is expected patients with more AEs are much more likely to discontinue treatment, more AEs tent to lead to higher medication non-adherence.
Adverse events affecting medication adherence | Month 3
  Secondary aim is to explore how adverse events (AE) impact medication adherence. AEs will be gathered throughout the duration of the study, assessed per seriousness, severity, causality and expectancy and descriptively presented. it is expected patients with more AEs are much more likely to discontinue treatment, more AEs tent to lead to higher medication non-adherence.
Adverse events affecting medication adherence | Month 6
  Secondary aim is to explore how adverse events (AE) impact medication adherence. AEs will be gathered throughout the duration of the study, assessed per seriousness, severity, causality and expectancy and descriptively presented. it is expected patients with more AEs are much more likely to discontinue treatment, more AEs tent to lead to higher medication non-adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Erika Matos, PhD, Principal Investigator — Institute of Oncology Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bray F, Laversanne M, Sung H, Ferlay J, Siegel RL, Soerjomataram I, Jemal A. Global cancer statistics 2022: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2024 May-Jun;74(3):229-263. doi: 10.3322/caac.21834. Epub 2024 Apr 4. PMID 38572751
- [Background] Siegel RL, Miller KD, Wagle NS, Jemal A. Cancer statistics, 2023. CA Cancer J Clin. 2023 Jan;73(1):17-48. doi: 10.3322/caac.21763. PMID 36633525
- [Background] Giaquinto AN, Sung H, Miller KD, Kramer JL, Newman LA, Minihan A, Jemal A, Siegel RL. Breast Cancer Statistics, 2022. CA Cancer J Clin. 2022 Nov;72(6):524-541. doi: 10.3322/caac.21754. Epub 2022 Oct 3. PMID 36190501
- [Background] Early Breast Cancer Trialists' Collaborative Group (EBCTCG). Aromatase inhibitors versus tamoxifen in early breast cancer: patient-level meta-analysis of the randomised trials. Lancet. 2015 Oct 3;386(10001):1341-1352. doi: 10.1016/S0140-6736(15)61074-1. Epub 2015 Jul 23. PMID 26211827
- [Background] Sheffield KM, Peachey JR, Method M, Grimes BR, Brown J, Saverno K, Sugihara T, Cui ZL, Lee KT. A real-world US study of recurrence risks using combined clinicopathological features in HR-positive, HER2-negative early breast cancer. Future Oncol. 2022 Jul;18(21):2667-2682. doi: 10.2217/fon-2022-0310. Epub 2022 May 25. PMID 35611679
- [Background] Gao JJ, Cheng J, Bloomquist E, Sanchez J, Wedam SB, Singh H, Amiri-Kordestani L, Ibrahim A, Sridhara R, Goldberg KB, Theoret MR, Kluetz PG, Blumenthal GM, Pazdur R, Beaver JA, Prowell TM. CDK4/6 inhibitor treatment for patients with hormone receptor-positive, HER2-negative, advanced or metastatic breast cancer: a US Food and Drug Administration pooled analysis. Lancet Oncol. 2020 Feb;21(2):250-260. doi: 10.1016/S1470-2045(19)30804-6. Epub 2019 Dec 16. PMID 31859246
- [Background] Johnston SRD, Harbeck N, Hegg R, Toi M, Martin M, Shao ZM, Zhang QY, Martinez Rodriguez JL, Campone M, Hamilton E, Sohn J, Guarneri V, Okada M, Boyle F, Neven P, Cortes J, Huober J, Wardley A, Tolaney SM, Cicin I, Smith IC, Frenzel M, Headley D, Wei R, San Antonio B, Hulstijn M, Cox J, O'Shaughnessy J, Rastogi P; monarchE Committee Members and Investigators. Abemaciclib Combined With Endocrine Therapy for the Adjuvant Treatment of HR+, HER2-, Node-Positive, High-Risk, Early Breast Cancer (monarchE). J Clin Oncol. 2020 Dec 1;38(34):3987-3998. doi: 10.1200/JCO.20.02514. Epub 2020 Sep 20. PMID 32954927
- [Background] Slamon D, Lipatov O, Nowecki Z, McAndrew N, Kukielka-Budny B, Stroyakovskiy D, Yardley DA, Huang CS, Fasching PA, Crown J, Bardia A, Chia S, Im SA, Ruiz-Borrego M, Loi S, Xu B, Hurvitz S, Barrios C, Untch M, Moroose R, Visco F, Afenjar K, Fresco R, Severin I, Ji Y, Ghaznawi F, Li Z, Zarate JP, Chakravartty A, Taran T, Hortobagyi G. Ribociclib plus Endocrine Therapy in Early Breast Cancer. N Engl J Med. 2024 Mar 21;390(12):1080-1091. doi: 10.1056/NEJMoa2305488. PMID 38507751
- [Background] Hershman DL, Shao T, Kushi LH, Buono D, Tsai WY, Fehrenbacher L, Kwan M, Gomez SL, Neugut AI. Early discontinuation and non-adherence to adjuvant hormonal therapy are associated with increased mortality in women with breast cancer. Breast Cancer Res Treat. 2011 Apr;126(2):529-37. doi: 10.1007/s10549-010-1132-4. Epub 2010 Aug 28. PMID 20803066
- [Background] Yussof I, Mohd Tahir NA, Hatah E, Mohamed Shah N. Factors influencing five-year adherence to adjuvant endocrine therapy in breast cancer patients: A systematic review. Breast. 2022 Apr;62:22-35. doi: 10.1016/j.breast.2022.01.012. Epub 2022 Jan 24. PMID 35121501
- [Background] Yeo HY, Liew AC, Chan SJ, Anwar M, Han CH, Marra CA. Understanding Patient Preferences Regarding the Important Determinants of Breast Cancer Treatment: A Narrative Scoping Review. Patient Prefer Adherence. 2023 Oct 31;17:2679-2706. doi: 10.2147/PPA.S432821. eCollection 2023. PMID 37927344
- [Background] Zhao M, Zhao J, Chen J, Li M, Zhang L, Luo X, Zhang Y, Xiong C, Guo Z, Yan J. The relationship between medication adherence and illness perception in breast cancer patients with adjuvant endocrine therapy: beliefs about medicines as mediators. Support Care Cancer. 2022 Dec;30(12):10009-10017. doi: 10.1007/s00520-022-07411-w. Epub 2022 Oct 20. PMID 36261611
- [Background] Agostinetto E, Vian L, Caparica R, Bruzzone M, Ceppi M, Lambertini M, Ponde N, de Azambuja E. CDK4/6 inhibitors as adjuvant treatment for hormone receptor-positive, HER2-negative early breast cancer: a systematic review and meta-analysis. ESMO Open. 2021 Apr;6(2):100091. doi: 10.1016/j.esmoop.2021.100091. Epub 2021 Mar 18. PMID 33743330
- [Background] Barroso-Sousa R, Shapiro GI, Tolaney SM. Clinical Development of the CDK4/6 Inhibitors Ribociclib and Abemaciclib in Breast Cancer. Breast Care (Basel). 2016 Jun;11(3):167-73. doi: 10.1159/000447284. Epub 2016 Jun 22. PMID 27493615
- [Background] Chan AHY, Horne R, Hankins M, Chisari C. The Medication Adherence Report Scale: A measurement tool for eliciting patients' reports of nonadherence. Br J Clin Pharmacol. 2020 Jul;86(7):1281-1288. doi: 10.1111/bcp.14193. Epub 2020 May 18. PMID 31823381
- [Background] Horne R, Weinman J. Patients' beliefs about prescribed medicines and their role in adherence to treatment in chronic physical illness. J Psychosom Res. 1999 Dec;47(6):555-67. doi: 10.1016/s0022-3999(99)00057-4. PMID 10661603
- [Background] Wagner L, Sweet J, Butt Z, Lai J, Cella D. Measuring patient self-reported cognitive function: development of the functional assessment of cancer therapy-cognitive function instrument. J Support Oncol. 2009;7(6):W32-9.
- [Background] Sprangers MA, Groenvold M, Arraras JI, Franklin J, te Velde A, Muller M, Franzini L, Williams A, de Haes HC, Hopwood P, Cull A, Aaronson NK. The European Organization for Research and Treatment of Cancer breast cancer-specific quality-of-life questionnaire module: first results from a three-country field study. J Clin Oncol. 1996 Oct;14(10):2756-68. doi: 10.1200/JCO.1996.14.10.2756. PMID 8874337
- [Background] Giesinger JM, Kieffer JM, Fayers PM, Groenvold M, Petersen MA, Scott NW, Sprangers MA, Velikova G, Aaronson NK; EORTC Quality of Life Group. Replication and validation of higher order models demonstrated that a summary score for the EORTC QLQ-C30 is robust. J Clin Epidemiol. 2016 Jan;69:79-88. doi: 10.1016/j.jclinepi.2015.08.007. Epub 2015 Sep 28. PMID 26327487
- [Background] Cancer EOfRaTo. Brussels: EORTC Brussels; 2001. Jan 01, Scoring of the QLQ-C30 Summary Score.
- [Background] Osoba D, Rodrigues G, Myles J, Zee B, Pater J. Interpreting the significance of changes in health-related quality-of-life scores. J Clin Oncol. 1998 Jan;16(1):139-44. doi: 10.1200/JCO.1998.16.1.139. PMID 9440735
- [Background] Bakovic M, Bago M, Benic L, Krajinovic M, Silovski T, Plavetic ND, Turkovic L, Sertic M, Hadziabdic MO. Exploring adherence in patients with advanced breast cancer: focus on CDK4/6 inhibitors. Acta Pharm. 2023 Dec 26;73(4):633-654. doi: 10.2478/acph-2023-0045. Print 2023 Dec 1. PMID 38147481
- [Background] Loucks J, Zuckerman AD, Berni A, Saulles A, Thomas G, Alonzo A. Proportion of days covered as a measure of medication adherence. Am J Health Syst Pharm. 2022 Mar 7;79(6):492-496. doi: 10.1093/ajhp/zxab392. No abstract available. PMID 34637496
- [Background] Burnier M. Is There a Threshold for Medication Adherence? Lessons Learnt From Electronic Monitoring of Drug Adherence. Front Pharmacol. 2019 Jan 9;9:1540. doi: 10.3389/fphar.2018.01540. eCollection 2018. PMID 30687099
- [Background] Yang S, Park SW, Bae SJ, Ahn SG, Jeong J, Park K. Investigation of Factors Affecting Adherence to Adjuvant Hormone Therapy in Early-Stage Breast Cancer Patients: A Comprehensive Systematic Review. J Breast Cancer. 2023 Aug;26(4):309-333. doi: 10.4048/jbc.2023.26.e22. Epub 2023 May 10. PMID 37272247
- See also: SmPC abemaciclib — https://www.ema.europa.eu/en/medicines/human/EPAR/verzenios
- See also: U.S Food and Drug Administration. FDA expands early breast cancer indication for abemaciclib with endocrine therapy 2023 — https://www.fda.gov/drugs/resources-information-approved-drugs/fda-disco-burst-edition-fda-approval-verzenio-abemaciclib-endocrine-therapy-patients-hr-positive
- See also: FACIT Group. FACT-Cog Scoring document — https://www.facit.org/measures/fact-cog
- See also: Fayers P, Bjordal K, Groenvold M, Curran D, Bottomley A. Brussels ORTC. Brussels: EORTC Brussels; 2001. EORTC QLQ-C30 Scoring Manual. 3rd ed. — https://www.eortc.org/app/uploads/sites/2/2018/02/SCmanual.pdf